CLINICAL TRIAL: NCT02746588
Title: Description of the Uterine Cavity in Patients With Recurrent Miscarriages
Status: Completed | Type: Observational
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Kristine Juul Hare, MD, PhD, Hvidovre University Hospital
Other Study IDs: H-15011157
Record Dates: First submitted 2016-04-18; First posted 2016-04-21 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Recurrent Miscarriages; Habitual Abortions
Keywords: miscarriage; uterine abnormalities; Chronic infection
MeSH Terms: conditions — Abortion, Habitual; Abortion, Spontaneous; Uterine Anomalies; Persistent Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Two endometrial biopsies
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Office hysteroscopy — Diagnostic hysteroscopy with biopsy

SUMMARY:
To be diagnosed with recurrent miscarriages, a couple might have a child, however experiences three or more miscarriages, primarily this happens during the first trimester.

These miscarriages often needs medical evacuation or a D & C. Surgery or retained tissue increases the risk of complications as infection and/or adhesions, known as asherman syndrome, which may result in subfertility.

Recently chronic infection in the endometrium has been proposed to contribute to the condition, as protocols including treatment with antibiotics have led to birth at term for some of these women.

Using the very minimal invasive office hysteroscopy, the investigators aim to describe the uterine cavity in patients diagnosed with recurrent miscarriages regarding both abnormalities in the endometrium and chromic infection.

DETAILED DESCRIPTION:
The Unit for Recurrent Pregnancy-loss at Rigshospitalet treats about 300 of couples with recurrent miscarriages a year. Together with the current examination program, the investigators plan to describe the uterine cavity according to abnormalities as septa, adhesions and further the condition for the endometrium regarding infection and hormone receptors. This description will include descriptive office hysteroscopy with biopsies for histologic - and immunohistochemically examinations.

ELIGIBILITY:
Inclusion Criteria:

* Correctly diagnosed with recurrent miscarriages

Exclusion Criteria:

* Known course of the condition

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients diagnosed with recurrent miscarriages and refurred to the specialist facility af Rigshospitalet
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Description of the Uterine Cavity in Patients With Recurrent Miscarriages | 1 year
  Observational study describing the uterine cavity in a selected patient group regarding abnormalities
Description of the Uterine Cavity in Patients With Recurrent Miscarriages | 1 year
  Observational study describing the uterine cavity in a selected patient group regarding chronic infection

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre Hospital, Department of Gynecology and Obstetrics, Copenhagen, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No